CLINICAL TRIAL: NCT02958423
Title: Transcranial Direct Current Stimulation (tDCS) vs Trans-spinal Direct Current Stimulation (tsDCS) for Endometriosis-related Chronic Pelvic Pain Treatment: A Single Center, Prospective, Randomized, Controlled, Parallel Group Pilot Study
Brief Title: tDCS Versus tsDCS for Endometriosis-related Chronic Pelvic Pain Treatment
Acronym: DCSErCPP
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jean Schoenen (Other)
Responsible Party: Sponsor-Investigator, Jean Schoenen, Professor, University of Liege
Organization: University of Liege (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B412201524615
Record Dates: First submitted 2016-11-01; First posted 2016-11-08 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Endometriosis; Pelvic Pain; Transcranial Direct Current Stimulation; Spinal Cord Stimulation
MeSH Terms: conditions — Endometriosis; Pelvic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Transcranial DCS Healthy Volunteers (Experimental): 5 HV will be treated once with transcranial direct current stimulation (2mA, anodal, 20 minutes) over right primary motor cortex with the Direct Current (DC) Stimulator (NeuroConn. Germany)
  Interventions: Device: Transcranial DCS Healthy Volunteers
- Transspinal DCS Healthy Volunteers (Experimental): 5 HV will be treated once with transspinal direct current stimulation (2mA, anodal, 20 minutes) over the D10 spinal process with the Direct Current (DC) Stimulator (NeuroConn. Germany)
  Interventions: Device: Transspinal DCS Healthy Volunteers
- Transcranial DCS CPP patients (Experimental): 5 chronic pelvic pain patients will be treated with transcranial direct current stimulation (2mA, anodal, 20 minutes) over right primary motor cortex 5 days/week for 4 weeks with the Direct Current (DC) Stimulator (NeuroConn. Germany)
  Interventions: Device: Transcranial DCS CPP patients
- Transspinal DCS CPP patients (Experimental): 5 chronic pelvic pain patients will be treated with transspinal direct current stimulation (2mA, anodal, 20 minutes) over the D10 spinal process 5 days/week for 4 weeks with the Direct Current (DC) Stimulator (NeuroConn. Germany)
  Interventions: Device: Transspinal DCS CPP patients

INTERVENTIONS:
Device: Transcranial DCS Healthy Volunteers — The DC stimulator manufactured by NeuroConn (Germany) will be used to deliver anodal direct current stimulation over the right primary motor cortex of healthy volunteers
  Arms: Transcranial DCS Healthy Volunteers
Device: Transspinal DCS Healthy Volunteers — The DC stimulator manufactured by NeuroConn (Germany) will be used to deliver anodal direct current stimulation over the D10 spinal process of healthy volunteers
  Arms: Transspinal DCS Healthy Volunteers
Device: Transcranial DCS CPP patients — The DC stimulator manufactured by NeuroConn (Germany) will be used to deliver anodal direct current stimulation over the right primary motor cortex of CPP patients
  Arms: Transcranial DCS CPP patients
Device: Transspinal DCS CPP patients — The DC stimulator manufactured by NeuroConn (Germany) will be used to deliver anodal direct current stimulation over the D10 spinal process of CPP patients
  Arms: Transspinal DCS CPP patients

SUMMARY:
The purpose of the study is to compare the analgesic effect of 2 mA anodal direct current stimulation on the right primary motor cortex (M1) (tDCS) with a similar stimulation on the spine (D10) (tsDCS) in healthy volunteers (HV) followed by a pilot study in patients suffering of endometriosis-related chronic pelvic pain (CPP)

DETAILED DESCRIPTION:
- 2 groups of 5 HV will receive tDCS or tsDCS (2mA, anodal, 20min) and the thermonociceptive threshold will be measured before and after the stimulation over the abdomen (hypogastric). The HAD scale and SF-36 will also be tested.

The treatment(s) that produces the greatest increase in pain thresholds will be chosen to treat 10 patients.

- 10 patients suffering from endometriosis-related chronic pelvic pain will be treated by the most efficient treatment (tDCS or tsDCS) for 4 weeks (5 daily 20-min sessions per week), or, if no treatment modality was superior in HV, 5 patients will be treated by tDCS and 5 by tsDCS. Patients will fill in daily a dedicated diary 2 weeks before treatment, during the4-week treatment period and after this period as long as their pain level remains below 80% of their baseline pain intensity (VAS). Analgesic intake will also be monitored as well as HAD and SF-36 scores.

ELIGIBILITY:
Inclusion Criteria:

* HV: good health.
* CPP patients: surgical diagnosis of endometriosis within the last 10 years; diagnosis of chronic pelvic pain (according to ACOG); mean VAS pain score >4 during severe episodes.

Exclusion Criteria:

* HV: chronic pain disorder; no regular medication or illicit drug use.
* CPP patients: pregnancy; other medical or psychiatric condition interfering with pelvic pain assessment.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-11 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Antalgic effect of direct current stimulation by measuring Quantitative Sensory Testing (QST) | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Nisolle, Professor, Principal Investigator — University of Liege
Locations (1):
- Departments of Gynecology & Neurology. CHR Citadelle, Liège, Belgium

IPD SHARING:
Plan to Share IPD: Yes
anonymized data will be made available on request via e-mail